CLINICAL TRIAL: NCT03122834
Title: Effect of Genetic Polymorphism on the Clinical Outcome, Echocardiographic Parameters and Cardiac Biomarkers of Patients With Heart Failure
Brief Title: Effect of Genetic Polymorphism on the Clinical Outcome of Patients With Heart Failure
Acronym: SNPs
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other); National Heart Institute (Unknown)
Responsible Party: Principal Investigator, Neven Sarhan, Lecturer of Clinical Pharmacy, Misr International University
Other Study IDs: SGLT2i-MRAs-ARNI
Record Dates: First submitted 2017-04-14; First posted 2017-04-21 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Genetic Polymorphism; RAAS; Cardiac Fibrosis; Remodeling
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected and stored in - 20°C environment for DNA extraction by DNA extraction kit according to manufacturer recommendation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: Newly diagnosed Heart Failure patients who will be treated with beta blockers (BB) and Angiotensin converting enzyme inhibitors (ACEIs)/or Angiotensin receptor blockers (ARBs) /or Angiotensin receptor neprilysin inhibitors (ARNI) and sodium glucose transporter 2 inhibitor (SGLT2i) for the first time.
- Cohort B: Heart Failure patients who are candidate for add-on treatment with Spironolactone / Eplerenone.

SUMMARY:
Heart failure (HF) is one the most common cause of hospitalization and represents the end stage of a variety of heart conditions; it is associated with significant morbidity and mortality.The pathophysiology of HF is centered on increased activity in the adrenergic and renin-angiotensin-aldosterone systems (RAAS), which leads to vasoconstriction and fluid restriction with further deleterious effect on cardiac function. Β-blockers, angiotensin converting enzyme inhibitors (ACEIs)/angiotensin II receptor blockers (ARBs) and aldosterone antagonists reduce activity in these pathways and have shown prognostic benefit, thus are the foundation of HF therapy.There is a growing body of evidence that variation in proteins within the sympathetic axis and RAAS influence drug response thus increasingly pharmacogenetics of HF research is being sought as a way to optimize HF treatment and advance new drug development in this area.

DETAILED DESCRIPTION:
In the past decade there has been considerable progress in cardiovascular pharmacogenetics and pharmacogenomics. Although drug response variation in Heart Failure is likely multifactorial, pharmacogenetic variation may partially account for therapeutic failure contributing to the remaining high mortality in HF. Identifying novel gene variants affecting treatment response may reveal unrecognized pathways and new potential therapeutic targets. Few studies to date have attempted to assess the extent to which variation in drug response was exclusively due to genetic factors and therefore expounding the likely clinical benefit of using pharmacogenetics to guide HF therapy. One of the prerequisites to bridging this gap is to consider likely trial designs and criteria that will lead to a consensus upon using pharmacogenetics-based variants to guide therapy in clinical practice.

Another area gaining momentum is tailoring medication in response to biomarker levels as there is considerable evidence for the relationship between remodeling and fibrosis markers levels and worse prognosis in those with HF. Moreover,investigation into the proteomics of HF may also reveal variation that can be used to guide HF therapy hand-in-hand with biomarkers and pharmacogenomics, which would facilitate bridging the gap of genotype and phenotype. Disparity between genotype and phenotype may also account for the inconsistent results with current SNPs, further appreciation of this relationship would be a significant step forward.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients NYHA class II to IV.
* Left ventricular ejection fraction (LVEF) < 45%
* Written informed consent of the subject to participate in the study.
* Newly diagnosed patients who will be treated with BBs and ACEIs/or ARBs.
* Patients who are candidate for add-on treatment with Spironolactone / Eplerenone.
* Age of 18 years to 80 years.

Exclusion Criteria:

* Contraindication to SGLT2i.
* Contraindication to Spironolactone / Eplerenone.
* Patients who received previous treatment with Spironolactone / Eplerenone.
* Sig CAD, CABG, PCI, or valve surgery within 3 months.
* Mild-to-severe valvular stenosis or severe (grade III/IV) valvular regurgitation
* Pregnant or nursing women.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Heart Failure Patients with reduced Ejection Fraction
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
RAAS genes and Clinical Outcome | 6 months
  Association between RAAS genetic polymorphism and clinical response, in-terms of change in LVEF among patients with heart failure
Adrenergic receptors genes and Clinical Outcome | 6 months
  Association between Adrenergic receptors genetic polymorphism and clinical response in terms of change in LVEF among patients with heart failure.
Cardiac Fibrosis genes and Clinical Outcome | 6 months
  Association between Cardiac Fibrosis genes genetic polymorphism and clinical response in terms of change in LVEF among patients with heart failure.
Reno-protective effect and gene polymorphism | 6 months
  Association between genetic polymorphism in SLC5A2, UMOD and ACE and Renal response in-terms of change in GFR among patients with heart failure.
RAAS genes and Biomarkers | 6 months
  Association between RAAS genetic polymorphism and Cardiac biomarkers among patients with heart failure.
Adrenergic receptors genes and Biomarkers | 6 months
  Association between Adrenergic receptors genetic polymorphism and Cardiac biomarkers among patients with heart failure.
Cardiac Fibrosis genes and Clinical Outcome | 6 months
  Association between Cardiac Fibrosis genes genetic polymorphism and Cardiac biomarkers among patients with heart failure.
Other Gene polymorphisms and Renal biomarkers | 6 months
  Association between genetic polymorphism in SLC5A2, UMOD and ACE and Renal biomarkers among patients with heart failure.

SECONDARY OUTCOMES:
Patients' mortality | 12 months
  Potential interaction between these target genes polymorphism and the 1 Year patients' mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Neven M. Sarhan, PhD, Principal Investigator — Misr International University; Mona F. Schaalan, PhD, Study Director — Misr International University; Bassem Zarif, MD, Study Chair — National Heart Institute
Locations (1):
- National Heart Institute, Cairo, Egypt